CLINICAL TRIAL: NCT03414931
Title: NMDA Modulation in Major Depressive Disorder in Late- Life
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101-0365A3
Record Dates: First submitted 2018-01-16; First posted 2018-01-30 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — N-Methylaspartate; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDA
- SSRI (Active Comparator): Sertraline
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: NMDA — Use of an NMDA enhancer for the treatment of MDD in late life
  Other Names: NMDAE
  Arms: NMDAE
Drug: Sertraline — Use of SSRI as an active comparator
  Arms: SSRI
Drug: Placebo - Cap — Use of placebo as a comparator
  Arms: Placebo

SUMMARY:
Major depressive disorder (MDD) is a complex and multi-factorial disorder. Most of the current antidepressants are based upon the monoamine hypothesis which cannot fully explain the etiology of depression. Many elderly patients have significant side effects after treatment with antidepressants which hamper the motivation for treatment and medication adherence. NMDA hypofunction has been implicated in the pathophysiology of depression. MDD in the elderly is often associated with cognitive deficits which are not necessarily recovered by current antidepressants. The NMDA receptor regulates synaptic plasticity, memory, and cognition. In our previous studies, cognitive improvement has been observed with treatment of NMDA enhancers. Therefore, this study will examine the efficacy and safety as well as cognitive function improvement of NMDAE in the treatment of MDD in the elderly by comparing with sertraline (a selective serotonin reuptake inhibitor [SSRI]) and placebo.

The investigator will enroll elderly patients with MDD for an 8-week treatment. All patients will be randomly assigned into three groups: NMDAE, sertraline, or placebo. The investigator will biweekly measure clinical performances. Cognitive functions will be assessed at baseline and at endpoint of treatment by a battery of tests. The investigator hypothesize that NMDAE can safely yield better efficacy than placebo and sertraline for elderly patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-IV (American Psychiatric Association 1994) diagnosis of MDD
* 17-item Hamilton Rating Scale for Depression total score ≥ 18
* Free of psychotropic drugs for at least 2 weeks
* Have a Mini-Mental State Examination (Folstein, Folstein et al. 1975) score ≥ 20

Exclusion Criteria:

* Current substance abuse or history of substance dependence in the past 6 months
* Use of depot antipsychotics in the past 6 months
* History of epilepsy, head trauma, stroke or other serious medical or neurological illness
* Bipolar depression, schizophrenia or other psychotic disorder
* Moderate-severe suicidal risks
* Severe cognitive impairment
* Initiating or stopping formal psychotherapy within six weeks prior to enrollment
* A history of poor response to SSRIs or other antidepressants
* A history of previously received electroconvulsive therapy
* A history of severe adverse reaction to SSRIs or other antidepressants
* Inability to follow protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of 17-item Hamilton Rating Scale for Depression | Week 0, 2, 4, 6, 8
  Assessment of depressive symptoms. The 17-item Hamilton Rating Scale for Depression will be measured biweekly.
Change from baseline of Perceived Stress Scale | Week 0, 2, 4, 6, 8
  Assessment of stress and anxiety symptoms. The Perceived Stress Scale will be measured biweekly

SECONDARY OUTCOMES:
Drop out rate | Week 0, 2, 4, 6, 8
  The rate of drop out
Change from baseline of Geriatric Depression Scale | Week 0, 2, 4, 6, 8
  Assessment of geriatric depressive symptoms. The Geriatric Depression Scale will be measured biweekly
Clinical Global Impression | Week 2, 4, 6, 8
  Assessment of global improvement
Cognitive function | Week 0, 8
  A battery of tests to assess the cognitive function including speed of processing (category fluency) and verbal and nonverbal working memory
Change from baseline of Beck's Suicide Scale | Week 0, 2, 4, 6, 8
  Assessment of suicidal symptoms. The Beck's Suicide Scale will be measured biweekly

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung

REFERENCES:
- [Derived] Lin CH, Wang SH, Lane HY. Effects of Sodium Benzoate, a D-Amino Acid Oxidase Inhibitor, on Perceived Stress and Cognitive Function Among Patients With Late-Life Depression: A Randomized, Double-Blind, Sertraline- and Placebo-Controlled Trial. Int J Neuropsychopharmacol. 2022 Aug 4;25(7):545-555. doi: 10.1093/ijnp/pyac006. PMID 35023557